CLINICAL TRIAL: NCT05073510
Title: A Prospective, Multicenter, Nonrandomized, Open-label, Single-arm Study of the BlueDop Vascular Expert for Assessing Peripheral Arterial Disease
Brief Title: Clinical Evaluation of the BlueDop Vascular Expert for Assessing Peripheral Arterial Disease
Status: Completed | Type: Observational
Sponsor: BlueDop Medical LTD (Industry)
Collaborators: AKRN Scientific Consulting, S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: BVE-01
Record Dates: First submitted 2021-09-15; First posted 2021-10-11 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; PAD; Arterial duplex
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BlueDop Vascular Expert (BVE): PAD assessment with BVE
  Interventions: Device: BVE

INTERVENTIONS:
Device: BVE — Participants will undergo BVE evaluation for assessing Peripheral Arterial Disease (PAD)

SUMMARY:
This is a BlueDop Vascular Expert System (BVE) Post-Market Clinical Follow-Up (PMCF) study. The primary objective of the study is to assess the clinical applicability and diagnostic accuracy of the BVE device in subjects who require an arterial duplex test due to suspected peripheral arterial disease (PAD).

DETAILED DESCRIPTION:
The BVE device is intended to assess mean peripheral pressure, vascular reserve, Cuff free Ankle Brachial Index (ABIm), and assess the presence or absence of hemodynamically significant arterial disease. By converting Doppler shifts to a blood pressure measurement, BVE can be used to monitor PAD in a non-invasive manner without confounding by arterial calcification.

This is a post-market, interventional, prospective, multi-center, open-label, non-randomized, single-arm clinical investigation designed to evaluate the clinical equivalence of BVE to arterial Duplex in a group of patients referred for evaluation of PAD of the limbs when performed by a vascular specialist. Moreover, the evaluation of the clinical performance including inter-operator variability and BVE non-diagnostic rate will be also carried out as exploratory variables.

1. Primary objective:

   Evaluate the clinical equivalence (assessment of accuracy) of BVE as binary result (either presence or absence of significant peripheral arterial disease) compared to arterial duplex ultrasound in a group of patients referred for evaluation of PAD of the lower limbs when performed by a vascular specialist.
2. Secondary objectives:

   Evaluate the clinical equivalence (assessment of accuracy) of BVE as binary result (either presence or absence of significant peripheral arterial disease) compared to ankle brachial pressure index (ABPI) in a group of patients referred for evaluation of PAD of the lower limbs when performed by a vascular specialist.

   Assess the safety of the BVE device.
3. Exploratory objectives:

Evaluation of the BVE System for clinical performance including time needed to perform BVE, inter-operator variability and number of BVE non-diagnostic tests.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent prior to any clinical investigation related procedure.
2. At least 18 years of age.
3. Referred for duplex ultrasound of the lower limb (s) with suspected or previous history of peripheral arterial disease
4. Must have an ABPI performed as part of the assessment
5. Able to obtain a brachial cuff blood pressure reading
6. Must have a valid ankle duplex ultrasound measurement at the Posterior Tibial Artery (PTA) and Dorsalis Pedis Artery (DPA)

Exclusion Criteria:

1. Subject is currently participating in another clinical investigation or has participated in another clinical investigation in the past 30 days prior to the start of the present study;
2. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period
3. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness;
4. Inability or refusal to give informed consent
5. Lower extremity wound or compromised skin of the legs that prevents access to the studied arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred for evaluation of PAD of the limbs when performed with duplex by a vascular specialist
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José Ignacio Leal Lorenzo, Principal Investigator — Clínica Universidad de Navarra
Locations (4):
- Spain (4):
  - Hospital Los Madroños, Brunete, Madrid
  - Hospital de Manises, Manises, Valencia
  - Clínica Universidad de Navarra, Madrid
  - Hospital Doctor Peset, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BlueDop Vascular Expert (BVE)
Started | 187
Completed | 186
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | BlueDop Vascular Expert (BVE)
Number analyzed (Participants) | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.24 (12.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 123
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 187

OUTCOME MEASURES:

1. Primary Outcome: Determination of Presence or Absence of Significant PAD With BVE and Arterial Duplex
Description: Evaluation of clinical equivalence through a binary result (either presence or absence of significant PAD) in BVE compared to a binary summary of the arterial duplex.
  Significant PAD is established with Duplex ultrasound when peak systolic velocity ratio (PSVR) is greater than 3 for any one level, or, if patients have multi-level disease, PSVR ≥ 2 at more than one level (i.e. sfa, pop)
Time Frame: 1 day
Population: ElP
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | BlueDop Vascular Expert (BVE)
Number analyzed (Participants) | 176
Number analyzed (Limbs) | 331
Limbs
  True Positives | 62
  False Positives | 14
  True Negatives | 212
  False Negatives | 43

2. Secondary Outcome: Determination of Presence or Absence of Significant PAD With BVE and ABPI
Description: Evaluation of clinical equivalence through a binary result (either presence or absence of significant PAD) in BVE compared to a binary summary of ABPI.
  Significant PAD is established when ABPI index is <0.8.
Time Frame: 1 day
Population: ElP
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | BlueDop Vascular Expert (BVE)
Number analyzed (Participants) | 176
Number analyzed (Limbs) | 326
Limbs
  True Positives | 62
  False Positives | 11
  True Negatives | 202
  False Negatives | 51

3. Secondary Outcome: Number and Risk-classification of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Evaluation of BVE safety through the assessment of the risk and occurrence rates of AEs and SAEs
Time Frame: 1 day
Measure: Number; unit: adverse events
Arm/Group | BlueDop Vascular Expert (BVE)
Number analyzed (Participants) | 187
adverse events | 0

4. Other Pre Specified Outcome: Time Spent for Arterial Duplex, BVE and ABPI Vascular Assessment
Description: Comparison of the time to perform a vascular assessment using arterial duplex, BVE, and ABPI (when available).
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- ABPI Time Cuff or Doppler: PAD assessment with ABPI Time cuff or doppler
- Duplex: PAD assessment with Duplex
- BVE-01: PAD assessment with BVE-01
- ABPI Automated Measure: PAD assessment with ABPI Automated measure
Arm/Group | ABPI Time Cuff or Doppler | Duplex | BVE-01 | ABPI Automated Measure
Number analyzed (Participants) | 187 | 187 | 187 | 187
minutes | 11.36 (6.14) | 16.90 (6.57) | 15.21 (11.24) | 11.39 (3.35)

5. Other Pre Specified Outcome: Determination of Presence or Absence of Significant PAD With BVE by Vascular and Non-vascular Experts
Description: Evaluation of clinical equivalence of BVE testing performed by staff specifically trained on BVE who are not vascular technologists/specialists compared to BVE testing performed by vascular technologists/specialists.
Time Frame: 1 day
Measure: Number; unit: Proportion of cases with agreement
Units Other Than Participants: Limbs
Groups:
- Vascular Expert vs Non-Vascular Expert PAD Assessment: PAD assessment with BVE by a Vascular Expert vs Non-Vascular Expert
Arm/Group | Vascular Expert vs Non-Vascular Expert PAD Assessment
Number analyzed (Participants) | 48
Number analyzed (Limbs) | 90
Proportion of cases with agreement | 0.8798

6. Other Pre Specified Outcome: BVE Non-diagnostic Rate
Description: Number of patients and/or limbs that could not be assessed by BVE.
Time Frame: 1 day
Population: This outcome was analyzed in the Enrollment population, not in the Eligible Population. The Eligible Population comprises the subset of enrolled patients who have at least one valid determination of PAD with both devices, and a limb without a valid PAD determination is considered analyzed if the other limb has a valid PAD determination. In the Enrollment Population we can find patients without any valid determination of PAD with BVE.
Measure: Count of Units; unit: Limbs
Units Other Than Participants: Limbs
Arm/Group | BlueDop Vascular Expert (BVE)
Number analyzed (Participants) | 187
Number analyzed (Limbs) | 353
Limbs | 74

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 day.
Arm/Group | BlueDop Vascular Expert (BVE)
All-Cause Mortality (participants affected / at risk) | 0/187
Serious Adverse Events (participants affected / at risk) | 0/187
Other Adverse Events (participants affected / at risk) | 0/187

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results and data obtained in the Clinical Trial shall be the exclusive property of the Sponsor, who reserves the right to use the results of this Trial to submit them to the authorities of any country.

DOCUMENTS (2):
  • Study Protocol (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT05073510/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT05073510/SAP_001.pdf